CLINICAL TRIAL: NCT03123848
Title: An Open-label Study to Evaluate the Pharmacokinetics (PK) of Darunavir (DRV) and Cobicistat (COBI) After a Single-oral Administration of Darunavir/Cobicistat Fixed-Dose Combination Tablet in Healthy Japanese Adult Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics (PK) of Darunavir (DRV) and Cobicistat (COBI) After a Single Oral Administration of Darunavir/Cobicistat Fixed-Dose Combination in Healthy Japanese Adult Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108319; TMC114FD1HTX4002 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2017-04-19; First posted 2017-04-21 (Actual); Results first posted 2018-06-12 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — cobicistat mixture with darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Darunavir/Cobicistat FDC (Prezcobix) (Experimental): Participants will receive one darunavir/cobicistat fixed-dose combination (FDC) tablet, containing 800 milligram (mg) of darunavir (DRV) and 150 mg of cobicistat (COBI) in the morning on Day 1.
  Interventions: Drug: Darunavir/Cobicistat

INTERVENTIONS:
Drug: Darunavir/Cobicistat — Participants will receive a FDC tablet of darunavir 800 mg and cobicistat 150 mg orally in the morning of Day 1.
  Other Names: TMC114/JNJ-48763364-AAA

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetic (PK) and safety of darunavir (DRV) and cobicistat (COBI) after a single oral administration of Prezcobix (DRV/COBI fixed-dose combination tablet) in healthy Japanese adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. This determination must be recorded in the participants source documents and initialed by the investigator
* A woman of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [hCG]) at screening and urine pregnancy test at the time of admission to the study site, hospitalization, and must not breast feed from screening onwards
* Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for participant participating in clinical studies
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of at least 30 days after intake of the study drug
* Nonsmoker or participant who habitually smokes no more than 10 cigarettes or equivalent of e-cigarettes, or 2 cigars, or 2 pipes of tobacco per day for at least 6 months before study drug administration

Exclusion Criteria:

* Participant has a history of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, liver or renal insufficiency (estimated creatinine clearance below 80 milliliter per minute [mL/min]); thyroid disease, neurologic or psychiatric disease, infection, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, metabolic disturbances or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Participant has a history of malignancy before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, that is considered cured with minimal risk of recurrence)
* Participant has a history of or current clinically significant skin reactions (such as but not limited to Stevens-Johnson Syndrome [SJS], Toxic Epidermal Necrolysis (TEN), and/or erythema multiforme) or any history of allergies to drugs, such as, but not limited to, sulfonamides and penicillins
* Participant has been contraindicated DRV and COBI per local prescribing information
* Participant is a woman, who is pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Souseikai Hakata Clinic, Fukuoka, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Darunavir 800 mg/Cobicistat 150 mg as FDC (Prezcobix): Participants received darunavir 800 milligram (mg) and Cobicistat 150 mg in a fixed-dose combination (FDC) as film-coated tablet formulation (PREZCOBIX) once orally on Day 1.
Period: Overall Study
Arm/Group | Darunavir 800 mg/Cobicistat 150 mg as FDC (Prezcobix)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Darunavir 800 mg/Cobicistat 150 mg as FDC (Prezcobix)
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (6.10)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8
Region of Enrollment [Count of Participants; unit: Participants]
  JAPAN | 8

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: The Cmax is the maximum observed plasma concentration.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 20, 24, 36, 48, 60, 72 hours postdose
Population: Pharmacokinetic (PK) analysis set included all participants who received the study drug and had at least one plasma concentration data-point after administration. Cmax for each analyte (Darunavir and Cobicistat) of fixed dose combination has been reported separately in each arm as per planned analysis.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Darunavir 800 mg (FDC: Darunavir 800/Cobicistat 150 mg); Cobicistat 150 mg (FDC: Darunavir 800/Cobicistat 150 mg): Participants received darunavir 800 mg along with cobicistat 150 mg in a fixed-dose combination (FDC) as film-coated tablet formulation (PREZCOBIX) once orally on Day 1.
Arm/Group | Darunavir 800 mg (FDC: Darunavir 800/Cobicistat 150 mg) | Cobicistat 150 mg (FDC: Darunavir 800/Cobicistat 150 mg)
Number analyzed (Participants) | 8 | 8
nanogram per milliliter (ng/mL) | 5496 (952) | 832 (265)

2. Primary Outcome: Concentration at Last Quantifiable Time Point (Clast)
Description: Clast is defined as concentration at last quantifiable time point.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 20, 24, 36, 48, 60, 72 hours postdose
Population: PK analysis set included all participants who received the study drug and had at least one plasma concentration data-point after administration. Clast for each analyte (Darunavir and Cobicistat) of fixed dose combination has been reported separately in each arm as per planned analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Darunavir 800 mg (FDC: Darunavir 800/Cobicistat 150 mg) | Cobicistat 150 mg (FDC: Darunavir 800/Cobicistat 150 mg)
Number analyzed (Participants) | 8 | 8
ng/mL | 33.3 (60.3) | 8.59 (3.24)

3. Primary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax)
Description: Tmax is defined as the time to reach the maximum plasma concentration.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 20, 24, 36, 48, 60, 72 hours postdose
Population: PK analysis set included all participants who received the study drug and had at least one plasma concentration data-point after administration. Tmax for each analyte (Darunavir and Cobicistat) of fixed dose combination has been reported separately in each arm as per planned analysis.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Darunavir 800 mg (FDC: Darunavir 800/Cobicistat 150 mg) | Cobicistat 150 mg (FDC: Darunavir 800/Cobicistat 150 mg)
Number analyzed (Participants) | 8 | 8
hour (h) | 4.00 [3.00 to 4.00] | 4.00 [2.00 to 4.00]

4. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Time the Last Quantifiable Time (AUC[0-last])
Description: AUC(0-last) is defined as area under the plasma concentration-time curve from time zero to time the last quantifiable time, calculated by linear trapezoidal summation.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 20, 24, 36, 48, 60, 72 hours postdose
Population: PK analysis set included all participants who received the study drug and had at least one plasma concentration data-point after administration time zero to time the last quantifiable time. AUC[0-last] for each analyte (Darunavir and Cobicistat) of fixed dose combination has been reported separately in each arm as per planned analysis.
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Darunavir 800 mg (FDC: Darunavir 800/Cobicistat 150 mg) | Cobicistat 150 mg (FDC: Darunavir 800/Cobicistat 150 mg)
Number analyzed (Participants) | 8 | 8
hour*nanogram per milliliter (h*ng/mL) | 51274 (15983) | 5667 (3119)

5. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC0-infinity)
Description: AUC(0-infinity) is defined as area under the plasma concentration-time curve from time zero to infinite time.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 20, 24, 36, 48, 60, 72 hours postdose
Population: PK analysis set included all participants who received the study drug and had at least one plasma concentration data-point after administration. AUC0-inf for each analyte (Darunavir and Cobicistat) of fixed dose combination has been reported separately in each arm as per planned analysis.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Darunavir 800 mg (FDC: Darunavir 800/Cobicistat 150 mg) | Cobicistat 150 mg (FDC: Darunavir 800/Cobicistat 150 mg)
Number analyzed (Participants) | 8 | 8
h*ng/mL | 51460 (15836) | 5710 (3128)

6. Primary Outcome: Elimination Rate Constant (Lambda[z])
Description: Lambda(z) is first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 20, 24, 36, 48, 60, 72 hours postdose
Population: PK analysis set included all participants who received the study drug and had at least one plasma concentration data-point after administration. Lambda[z] for each analyte (Darunavir and Cobicistat) of fixed dose combination has been reported separately in each arm as per planned analysis.
Measure: Mean (Standard Deviation); unit: per hour (1/h)
Arm/Group | Darunavir 800 mg (FDC: Darunavir 800/Cobicistat 150 mg) | Cobicistat 150 mg (FDC: Darunavir 800/Cobicistat 150 mg)
Number analyzed (Participants) | 8 | 8
per hour (1/h) | 0.173 (0.0668) | 0.199 (0.0233)

7. Primary Outcome: Terminal Elimination Half-Life (t1/2)
Description: t1/2 is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 20, 24, 36, 48, 60, 72 hours postdose
Population: PK analysis set included all participants who received the study drug and had at least one plasma concentration data-point after administration. t1/2 for each analyte (Darunavir and Cobicistat) of fixed dose combination has been reported separately in each arm as per planned analysis.
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Darunavir 800 mg (FDC: Darunavir 800/Cobicistat 150 mg) | Cobicistat 150 mg (FDC: Darunavir 800/Cobicistat 150 mg)
Number analyzed (Participants) | 8 | 8
Hour | 4.4 (1.4) | 3.5 (0.4)

8. Primary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Vz/F is defined as the apparent volume of distribution at the terminal phase after extravascular administration.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 20, 24, 36, 48, 60, 72 hours postdose
Population: PK analysis set included all participants who received the study drug and had at least one plasma concentration data-point after administration. Vz/F for each analyte (Darunavir and Cobicistat) of fixed dose combination has been reported separately in each arm as per planned analysis.
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Darunavir 800 mg (FDC: Darunavir 800/Cobicistat 150 mg) | Cobicistat 150 mg (FDC: Darunavir 800/Cobicistat 150 mg)
Number analyzed (Participants) | 8 | 8
milliliter (mL) | 111970 (61217) | 166460 (76366)

9. Primary Outcome: Apparent Total Body Clearance of Drug at the Terminal Phase After Extravascular Administration (CL/F)
Description: CL/F is the apparent total body clearance of drug at the terminal phase after extravascular administration.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 20, 24, 36, 48, 60, 72 hours postdose
Population: PK analysis set included all participants who received the study drug and had at least one plasma concentration data-point after administration. CL/F for each analyte (Darunavir and Cobicistat) of fixed dose combination has been reported separately in each arm as per planned analysis.
Measure: Mean (Standard Deviation); unit: milliliter per hour (mL/h)
Arm/Group | Darunavir 800 mg (FDC: Darunavir 800/Cobicistat 150 mg) | Cobicistat 150 mg (FDC: Darunavir 800/Cobicistat 150 mg)
Number analyzed (Participants) | 8 | 8
milliliter per hour (mL/h) | 16974 (5440) | 33573 (16699)

10. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Time Frame: Up to approximately 1 month
Population: Safety analysis set included all participants who received the study drug. AEs for each analyte (Darunavir and Cobicistat) of fixed dose combination has been reported separately as per planned analysis.
Measure: Number; unit: Participants
Arm/Group | Darunavir 800 mg/Cobicistat 150 mg as FDC (Prezcobix)
Number analyzed (Participants) | 8
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 1 month
Description: Safety analysis set included all participants who received the study drug.
Arm/Group | Darunavir 800 mg/Cobicistat 150 mg as FDC (Prezcobix)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-02-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT03123848/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT03123848/SAP_001.pdf